CLINICAL TRIAL: NCT01304966
Title: Human Papillomatosis Genotyping and Severity in Patients With Recurrent Respiratory Papillomatosis of Children in Thailand
Brief Title: Human Papillomatosis Genotyping of Children in Thailand
Status: Completed | Type: Observational
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Pavinee Intakorn, department of otorhinolarngology, Queen Sirikit National Institute of Child Health
Other Study IDs: qnischent01
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Laryngeal Papillomatosis; Human Papilloma Virus
Keywords: RRP; HPV
MeSH Terms: conditions — Laryngeal papillomatosis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Papillomatous tissue samples taken from endoscopic biopsies will be collected by the ENT specialists.Samples collected from the subjects will be analyzed for HPV genotype at the Unit of virology and molecular, Department of pathology, Faculty of medicine Ramathibodi hospital.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: biopsy — excisional biopsy

SUMMARY:
The purpose of the present study was to identify risk factors for more severe juvenile Recurrent Respiratory Papillomatosis (RRP) through prospective evaluation of a pediatric population in Thailand by the employing a protocol that includes staging of disease severity using above mentioned staging system at the time of each endoscopic debridement, as well as human papilloma virus (HPV) genotyping.

DETAILED DESCRIPTION:
Recurrent respiratory papillomatosis is caused by human papilloma virus and is the most common benign laryngeal neoplasm in children. Although RRP is rarely fatal, the disease requires prolonged, extensive medical and surgical treatment, and causes physical and emotional suffering in affected children and their families. Although recurrent respiratory papillomatosis is a relatively unusual problem, it accounts for significant health are expenditures.The goal of management of RRP is control of the disease, preservation of the voice and prevention of major complication .The purpose of study will identify risk factors for more severe juvenile RRP through prospective evaluation of a pediatric population in Thailand by the employing a protocol that includes staging of disease severity , as well as HPV genotyping.

Objective:

* To identify the genotypes of HPV isolated from Thai RRP patients
* To compare staging and severity with HPV genotypes
* To correlate the following characteristics of the Thai RRP patients with the HPV genotypes

ELIGIBILITY:
Inclusion Criteria:

* Patients have active laryngeal papillomatosis .
* Patients have developed this infection before the age of 18 years old.

Exclusion Criteria:

* Children whose families do not sign an informed consent to enter into study.
* Children whose families anticipate discontinuing care at a participating institution during the study period.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Target enrollment will be all children who are diagnosed with RRP.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavinee Intakorn, MD, Principal Investigator — Queen Sirikit National Institute of Child Health; Pavinee Intakorn, MD, Principal Investigator — Queen Sirikit National of Child Health
Locations (2):
- Thailand (2):
  - Department of Otorhinolaryngology: Queen Sirikit National of Child Health, Bangkok, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok, Bangkok

REFERENCES:
- [Background] Derkay CS. Task force on recurrent respiratory papillomas. A preliminary report. Arch Otolaryngol Head Neck Surg. 1995 Dec;121(12):1386-91. doi: 10.1001/archotol.1995.01890120044008. PMID 7488368
- [Background] Doyle DJ, Gianoli GJ, Espinola T, Miller RH. Recurrent respiratory papillomatosis: juvenile versus adult forms. Laryngoscope. 1994 May;104(5 Pt 1):523-7. doi: 10.1002/lary.5541040503. PMID 8189980
- [Background] Kashima HK, Shah F, Lyles A, Glackin R, Muhammad N, Turner L, Van Zandt S, Whitt S, Shah K. A comparison of risk factors in juvenile-onset and adult-onset recurrent respiratory papillomatosis. Laryngoscope. 1992 Jan;102(1):9-13. doi: 10.1288/00005537-199201000-00002. PMID 1309932
- [Background] Rabah R, Lancaster WD, Thomas R, Gregoire L. Human papillomavirus-11-associated recurrent respiratory papillomatosis is more aggressive than human papillomavirus-6-associated disease. Pediatr Dev Pathol. 2001 Jan-Feb;4(1):68-72. doi: 10.1007/s100240010105. PMID 11200493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of the recruitment is APril 2011.Number participants staring is fifteen.
Groups:
- Children With Recurrent Respiratory Papillomatosis: Children hospitalized with recurrent respiratory papillomatosis who underwent biopsy
Period: Overall Study
Arm/Group | Children With Recurrent Respiratory Papillomatosis
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children With Recurrent Respiratory Papillomatosis in Thailand
Arm/Group | Children With Recurrent Respiratory Papillomatosis
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.67 (0.049)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Human Papillomavirus Genotypes
Description: Distribution of Human papillomavirus(HPV) genotypes identified in the biopsy
Time Frame: 12 months
Population: We found positive HPV DNA in all children. HPV type 6 and HPV type 11 caused recurrent respiratory papillomatosis in 6 (40%) and 9(60%) of cases,respectively.
Measure: Number; unit: participants
Groups:
- Children With Recurrent Respiratory Papillomatosis: Distribution of Human papillomavirus(HPV) genotypes identified in the biopsy
Arm/Group | Children With Recurrent Respiratory Papillomatosis
Number analyzed (Participants) | 15
participants
  HPV type 6 | 6
  HPV type 11 | 9

2. Secondary Outcome: Cotreta-Derkay Score
Description: We compared disease severity(Cotreta-Derkay score) between groups of children with two different HPV genotypes
  Coltera and Derkay have evolved a staging system to stage recurrent papillomatous lesions involving the respiratory tract.
  Coltera-Derkay method of staging :
  Clinical score:
  1. Voice: Normal - 0, Abnormal - 1, Aphonia - 2
  2. Stridor: Absent - 0, Present on activity - 1, Present at rest - 2
  3. Respiratory distress - None - 0, Mild - 1, Moderate - 2, Severe - 3, Extreme - 4.
  Anatomical score:
  For each site - 0 = none, 1=surface lesion, 2= raised lesion, 3=bulky lesion.
  Total score = Anatomical score + Total clinical score
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score
Groups:
- HPV 6: Children with recurrent respiratory papillomatosis from HPV 6
- HPV 11: Children with recurrent respiratory papillomatosis from HPV 11
Arm/Group | HPV 6 | HPV 11
Number analyzed (Participants) | 6 | 9
score | 13.83 (9.94) | 27.44 (8.24)
Statistical Analysis 1: Comparison: HPV 6 vs HPV 11; Test type: Superiority or Other; p = 0.013, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 12 months
Description: Since this is the observational study, therefore the study process did not pose any risk to the participants (population at risk = 0)
Arm/Group | Children With Recurrent Respiratory Papillomatosis
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The number of patients participating in this study was low , so additional studies should be conducted to make the research more effective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes